CLINICAL TRIAL: NCT06624683
Title: Exploring the Effect of Footbaths on Increasing the Success Rates of in Vitro Fertilization and Its Associated Mechanism
Brief Title: Exploring the Effect of Footbaths on Increasing the Success Rates in Vitro Fertilization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, YA-WEN SHIH, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-06-009BC
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Infertility; In Vitro Fertilization
Keywords: Infertility; In vitro fertilization; Stress; Sleep quality; Inflammation; Footbath
MeSH Terms: conditions — Infertility; Sleep Initiation and Maintenance Disorders; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervation (Experimental): Participants in the intervention group will immerse their feet up to 10 cm into water inside a collapsible plastic container, maintaining a temperature of 40°C for 30 minutes every night, one hour before usual bedtime (between 21:00 and 22:00), starting from the first day of the menstrual cycle (MC) and continuing for 28 days.
  Interventions: Device: Intelligent footbath basin
- usual care (No Intervention): clinical usual care

INTERVENTIONS:
Device: Intelligent footbath basin — before night sleep, takes 30 mins, starting from the first day of the menstrual cycle (MC) and continuing for 28 days.
  Arms: intervation

SUMMARY:
To evaluate the effectiveness of warm-water footbaths in enhancing pregnancy rates during IVF and to explore the underlying mechanisms involved.

DETAILED DESCRIPTION:
Additionally, this research will assess whether a complementary and alternative medicine (CAM) approach utilizing warm-water footbaths is effective in improving pregnancy rates for women undergoing IVF. Furthermore, the potential mechanisms by which footbaths may enhance IVF success rates will be elucidated.

The specific aims of this research proposal are as follows:

1. To explore the correlation between health statuses, sleep quality, stress, and infertility incidence.
2. To investigate the association between health statuses, sleep quality, stress, and multiple inflammatory indexes in infertile women, including:

   2-1. Systemic immune inflammation index (SII) 2-2. Lymphocyte count (LC) 2-3. Platelet and neutrophil count product (PPN) 2-4. Platelet-lymphocyte ratio (PLR) 2-5. Neutrophil-lymphocyte ratio (NLR) 2-6. Lymphocyte-monocyte ratio (LMR)
3. The effects of Footbaths on Stress and Sleep:

   To examine the effects of footbaths on reducing stress and improving sleep quality, which may enhance pregnancy success rates during IVF treatment in infertile women.
4. The impact on Inflammatory Markers:

To investigate whether footbaths can reduce levels of inflammatory markers and inflammatory cytokines during IVF treatment, potentially enhancing pregnancy success rates in infertile women.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18~45 years
* diagnosed with male factor infertility
* tubal factor infertility, or unexplained infertility, and undergoing an IVF treatment.

Exclusion Criteria:

* participants having adenomyosis, severe endometriosis
* a history of more than two IVF treatments
* any comorbidity or uncontrolled systemic diseases such as hypertension, diabetes, chronic heart disease or chronic renal disease that can affect the treatment process.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 28 days
  IVF success rates in infertile women

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hong Ho, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No